CLINICAL TRIAL: NCT07032675
Title: Cartilage Remodeling Using Low-Temperature Radiofrequency for Facial Reconstruction
Brief Title: Cartilage Remodeling Using Low-Temperature Radiofrequency for Nasal Airway Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Taha Shipchandler, Division Chief of Facial Plastic and Reconstructive Surgery in the Department of Otolaryngology-Head and Neck Surgery, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24964
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Nasal Valve Collapse; Nose Enhancement
Keywords: low-temperature radio-frequency; nasal valve collapse; septorhinoplasty; septoplasty; rhinoplasty; cartilage reshaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low-temperature radio-frequency reshaping intervention (Experimental): All enrolled subjects will receive the intervention outlined in the section titled "Study Design".
  Interventions: Device: Low-temperature radio-frequency reshaping of autologous cartilage nasal and/or auricular cartilage

INTERVENTIONS:
Device: Low-temperature radio-frequency reshaping of autologous cartilage nasal and/or auricular cartilage — The device settings will be set per the manufacturer's instructions: temperature = 60° C, power = 4 W, treatment time = 18 seconds, and cooldown = 12 seconds. For curved-to-straight (CTS) samples (natively curved cartilage to be remolded to be flat), the cartilage specimens will be placed on a blue towel on a flat surface with the transmission medium over top and treated. For straight-to-curved (STC) samples (natively flat cartilage to be remolded to be curved), cartilage specimens will be placed along the inner surface of various shallow, plastic, cylindrical objects with the transmission medium over top and treated. Various device settings may be tested for reshaping efficacy.

SUMMARY:
The goal of this study is to evaluate the efficacy of using the Vivaer low-temperature radio-frequency (LTRF) device to reshape ex-vivo human nasal or auricular cartilage for use in cosmetic and functional septorhinoplasty. The investigators hope to answer the following questions:

1. How many LTRF treatments are needed to achieve the desired shape in a given cartilage specimen
2. How does an LTRF treatment quantitatively affect both length and angulation of a cartilage specimen
3. How does physician satisfaction with cosmetic outcome compare to cases treated with existing septorhinoplasty techniques
4. How do changes in patient reported measures of nasal obstruction (NOSE score) pre- and post-surgery compare to cases treated with existing septorhinoplasty techniques
5. Does using LTRF during septorhinoplasty significantly increase total operative time
6. Are rates of adverse events when using LTRF different from cases treated with existing septorhinoplasty techniques

Participants will complete the NOSE questionnaire at their pre-operative visit. Participants undergoing cosmetic septhorhinoplasty will also be photographed in standard fashion for facial analysis.

During scheduled septorhinoplasty surgery, the Vivaer LTRF device will be used to reshape nasal and/or auricular cartilage ex-vivo prior to reimplantation at the discretion of the Principal Investigator in order to optimize functional and cosmetic outcome.

Participants will follow up at approximately 1 week and 1 month after surgery. At 1 month, the NOSE questionnaire will be readministered to all participants, and cosmetic patients will be photographed again.

ELIGIBILITY:
Inclusion Criteria:

• Patients 18 years and older undergoing functional septorhinoplasty or cosmetic septorhinoplasty, with or without auricular cartilage harvest

Exclusion Criteria:

* Patients who have had a prior septorhinoplasty
* Patients who have received prior head and neck radiation
* Patients with a septal perforation
* Patients who are medically ineligible to undergo septorhinoplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of treatments needed to reach desired shape | Immediately pre and post intervention (intraoperative)
  The primary outcome measure will be the efficacy of reshaping cartilage from straight to curved and from curved to straight for use in septorhinoplasty. The number of treatments needed to create the desired shapes and curvatures will be measured for each cartilage specimen.

SECONDARY OUTCOMES:
Change in specimen curvature | Immediately pre and post intervention (intraoperative)
  The angle of curvature of each specimen will be measured as the angle of the intersection between two lines drawn along the distal edges of the specimen. The difference in angle of curvature before and after low-temperature radiofrequency treatment will be calculated.
Change in specimen length | Immediately pre and post intervention (intraoperative)
  The apparent length of each specimen before and after treatment will be measured as a straight line between the distal points of the cartilage sample. . The differences in length before and after low-temperature radiofrequency treatment will be calculated.
Nasal Obstruction Symptom Evaluation (NOSE) score | Baseline and one month
  Nasal Obstruction Symptom Evaluation (NOSE) score, a validated patient-reported outcome measure of nasal airway obstruction, will be obtained at the first pre-operative visit and at the second post-operative visit (approximately 1 month after surgery). Nasal obstruction severity classification: mild (5-25) moderate (30-50) severe (55-75) extreme (80-100).
Physician satisfaction with cosmetic outcome | Baseline and one month
  Preoperative and postoperative standard septorhinoplasty photographs will be compared and rated by the surgeon. In cosmetic rhinoplasty, it is standard practice to take full-face patient photographs before and after surgery to assess cosmetic outcomes (frontal, lateral, oblique, nasal base angles). Full face photographs are necessary to include all soft tissue and bony landmarks to assess nasal proportions relative to the face. They will be stored in the Vectra imaging suite software used for facial plastic surgery photography, which is currently in use clinically and is HIPPA-compliant.

OTHER OUTCOMES:
Reimplantation of LTRF-shaped specimens | Immediately pre and post intervention (intraoperative)
  Binary documentation of whether or not LTRF-shaped specimens are ultimately reimplanted.
Time spent using low-temperature radiofrequency device | Immediately pre and post intervention (intraoperative)
  Time spent (minutes) using LTRF device will be recorded to quantify addition of operative time.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - IU Health North Hospital, Indianapolis, Indiana
  - IU Health Saxony Hospital, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - IU Health West Hospital, Indianapolis, Indiana
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana